CLINICAL TRIAL: NCT01216865
Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cells Injection for Diabetic Foot
Brief Title: Umbilical Cord Mesenchymal Stem Cells Injection for Diabetic Foot
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Wang, Yangang MD, Stem Cell Research Center of Medical School Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSCDF001
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2009-01

CONDITIONS: Diabetic Foot; Critical Limb Ischemia; Mesenchymal Stem Cells; Umbilical Cord
Keywords: Diabetic foot; critical limb ischemia; mesenchymal stem cells; umbilical cord
MeSH Terms: conditions — Diabetic Foot; Chronic Limb-Threatening Ischemia | interventions — Standard of Care; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- umbilical cord mesenchymal stem cells (Experimental): Multiple intra muscular injection of mesenchymal stem cells derived from human umbilical cord.
  Interventions: Biological: umbilical cord mesenchymal stem cells
- Standard Therapy (Active Comparator): Any therapy for diabetic foot which is routinely practiced and accepted in China
  Interventions: Drug: Standard Therapy

INTERVENTIONS:
Biological: umbilical cord mesenchymal stem cells — 5*10/7 per ischemic limb
  Other Names: mesenchymal stem cells
  Arms: umbilical cord mesenchymal stem cells
Drug: Standard Therapy — Any thing directed to improve blood perfusion in the limb example.Heparin,Antiplatelet agents etc
  Other Names: Drug therapy
  Arms: Standard Therapy

SUMMARY:
The purpose of this study is to determine whether umbilical cord Mesenchymal Stem Cells of treatment for diabetic foot is safe and effective in the management of diabetic foot ischemia, the therapeutic effect of stem cells is caused by improving blood circulation in ischemic limb which would in turn promote ulcer healing, prevent amputation of limb and relieve the Sevier pain of ischemia.

DETAILED DESCRIPTION:
Type 2 diabetic patients with diabetic foot were enrolled and randomized to either transplanted group or control group. Patients in transplanted group received the stem cells treatment,Patients in control group received the standard treatment. After culture in vitro, umbilical cord mesenchymal stem cells should go through safety evaluation which include culture and check of pathogenic microorganisms (bacteria, mycoplasma, chlamydia, eumycete and viruses) of the cells medium and karyotype analysis of the mesenchymal stem cells. Only the safe cells were harvested and transplanted by multiple intramuscular injections into the impaired lower limbs. Follow-up index include: efficacy (pain,ulcer healing rate, lower limb amputation rate and ,ankle-brachial index,magnetic resonance angiography,electromyogram) and safety (infection of the injection site, fever, and tumour generation).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus Type 2
* Age 18 - 75 years
* Subject has an Ankle-brachial index < 0.9
* Subject has had previous conservative treatment which resulted in little or no improvement
* Subject has had no stem cell treatment within the past 6 months
* No sufficient response to best standard care delivered for six weeks.
* No surgical or radiological interventional option for revascularisation as confirmed by a vascular surgeon and an interventional radiologist
* Signed informed consent
* Absence of life-threatening complications from the ischemic limb
* Life expectancy more than 2 years
* Negative pregnancy test when applicable

Exclusion Criteria:

* Diabetic retinopathy
* History of neoplasm or hematological disease
* Uncontrolled high blood pressure (>180/110)
* Severe cardiac insufficiency (New York Heart Association [NYHA] IV) or ejection fraction<30%
* Malignant ventricular arrythmia
* Deep venous thrombosis during the last 3 months
* Active bacterial infection
* Body mass index > 35 Kg/m2
* Stroke or myocardial infarction during the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Angiographic evaluation of angiogenesis at ischemic limb | 6 months

SECONDARY OUTCOMES:
Pain | 3 months
Ankle-Brachial pressure index | 3 months
Wound healing (wound size, wound stage) | 3 months
Walking distance | 3 months
Rate and extent of amputations | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yangang Wang, MD Phd, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Stem Cell Research Center of Medical School Hospital of Qingdao University, Qingdao, Shandong, China